CLINICAL TRIAL: NCT04923399
Title: Transcriptome Sequencing Analysis of Whole Blood From Patients With Trigeminal Neuralgia: An Observational Study
Brief Title: Transcriptome Sequencing Analysis of Whole Blood From Patients With Trigeminal Neuralgia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Chief of the Anesthesiology Department, Peking University People's Hospital
Other Study IDs: 2020PHB265-01
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Trigeminal Neuralgia; Blood; Plasma; Cerebrospinal Fluid
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — whole blood cell; plasma; cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TN (Trigeminal Neuralgia) group: Trigeminal neuralgia patients undergoing trigeminal nerve microvascular decompression
- Non-TN group: patients without chronic pain or history of chronic pain

SUMMARY:
Trigeminal neuralgia is a type of neuropathic pain that brings great physical and psychological pressure to patients. Chronic pain can cause changes in the composition of central and peripheral body fluids, and these changes may be useful for the prediction and treatment of pain. In this study, the whole blood of patients with trigeminal neuralgia and non-chronic pain was collected, and transcriptome sequencing (RNA-seq) was performed to determine the peripheral transcriptome changes of trigeminal neuralgia (TN) patients. And compare the expression of neuropeptide Y (NPY) in plasma and cerebrospinal fluid of TN and non-chronic pain patients.

DETAILED DESCRIPTION:
Trigeminal neuralgia is a kind of paroxysmal, knife-cutting, stubborn and severe pain in the facial distribution area of the trigeminal nerve caused by slight stimulation, which brings a great physical and psychological burden to the patient. Chronic pain can cause changes in the composition of central and peripheral body fluids, and these changes are very useful for the prediction and treatment of pain. In this study, the whole blood of patients with trigeminal neuralgia and non-chronic pain was collected for transcriptome sequencing (RNA-seq) sequencing. The results of transcriptome sequencing can derive the differentially expressed genes in the whole blood of TN patients and the pathways enriched by differentially expressed genes. At the same time, NPY (Neuropeptide y) plays an important role in head and face pain. We will also verify the difference in NPY expression in the cerebrospinal fluid and plasma of TN and non-chronic pain patients, and the correlation between NPY expression and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary trigeminal neuralgia receive trigeminal nerve microvascular decompression, and healthy people without a history of chronic pain or patients with facial nerve palsy without chronic pain receive facial nerve decompression as a control;
2. Age from 30 to 60 years old
3. Complete white blood cell count: 4.8~11.0x109/L

Exclusion Criteria:

1. Patients with co-infection and tumor
2. Patients with craniocerebral disease

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Trigeminal neuralgia patients receive the trigeminal nerve microvascular decompression surgery. The comparsion group is patients without chronic pain or history of chronic pain. The whole blood cell, plasma and cerebrospinal fluid will be collected during the perioperative period.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | The VAS score is tested before surgery in the preoperative preparation room
  VAS score is a pain score
Differentially expressed genes | blood will be taken from two groups of patients before operation
  Transcriptome analysis of whole blood cell from patients with trigeminal neuralgia or non-chronic pain reveals differential gene expression between the two groups
Differentially expressed genes (DEGs) enrichment pathway | blood will be taken from two groups of patients before operation
  We will perform pathway enrichment analysis on the DEGs obtained by transcriptome analysis of the whole blood cell from patients with trigeminal neuralgia or non-chronic pain.
Neuropeptide y expression | Cerebrospinal fluid will be collected during the surgery; Plasma will be collected before the surgery in the preoperative preparation room.
  We detect neuropeptide Y levels in the cerebrospinal fluid and plasma of patients with trigeminal neuralgia and non-chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, PhD, Principal Investigator — Peking University People's Hospital

REFERENCES:
- [Background] Montano N, Conforti G, Di Bonaventura R, Meglio M, Fernandez E, Papacci F. Advances in diagnosis and treatment of trigeminal neuralgia. Ther Clin Risk Manag. 2015 Feb 24;11:289-99. doi: 10.2147/TCRM.S37592. eCollection 2015. PMID 25750533
- [Background] Song N, Liao DQ, Liu F, Zhang YY, Lin J, Wang H, Shen JF. Effect of Titanium Particles on the Voltage-Gated Potassium Channel Currents in Trigeminal Root Ganglion Neurons. Implant Dent. 2019 Feb;28(1):54-61. doi: 10.1097/ID.0000000000000848. PMID 30507652
- [Background] Eroli F, Loonen ICM, van den Maagdenberg AMJM, Tolner EA, Nistri A. Differential neuromodulatory role of endocannabinoids in the rodent trigeminal sensory ganglion and cerebral cortex relevant to pain processing. Neuropharmacology. 2018 Mar 15;131:39-50. doi: 10.1016/j.neuropharm.2017.12.013. Epub 2017 Dec 7. PMID 29225040
- [Derived] Liu T, Xu C, Guo J, He Z, Zhang Y, Feng Y. Whole Blood Transcriptome Analysis in Patients with Trigeminal Neuralgia: a Prospective Clinical Study. J Mol Neurosci. 2024 Feb 1;74(1):16. doi: 10.1007/s12031-024-02195-6. PMID 38300339